CLINICAL TRIAL: NCT03164330
Title: Illinois Workplace Wellness Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other); University of Chicago (Other); National Institutes of Health (NIH) (NIH); Robert Wood Johnson Foundation (Other); Abdul Latif Jameel Poverty Action Lab (Other); W.E. Upjohn Institute for Employment Research (Unknown); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Damon Jones, Faculty Research Fellow, National Bureau of Economic Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0008; R01AG050701 (NIH); 73730 (Other Grant/Funding Number: Robert Wood Johnson Foundation); 2016-06638 (Other Grant/Funding Number: Abdul Latif Jameel Poverty Action Lab)
Record Dates: First submitted 2017-05-17; First posted 2017-05-23 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Employee Health and Well-being
Keywords: Health Care; Workplace Wellness; Preventative Health Care; Health Costs
MeSH Terms: interventions — Risk Assessment

STUDY DESIGN:
Intervention Model Description: Our primary analysis compares outcomes between a control group and six (6) treatment groups. Our secondary analysis compares pre-determined characteristics across members of the treatment group who adopt the intervention and those who do not.
Who Masked: Care Provider
Masking Description: Professionals who implement the biometric screenings, health risk assessments, and wellness courses do no know the exact treatment group of study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control (No Intervention): The control group takes a baseline survey, and thereafter has minimal interaction with the project, until a follow-up biometric screening is conducted during the one-year follow-up.
- A25 (Experimental): Group A25 is offered no compensation for completing a biometric screening and HRA, and low compensation for each completed wellness course in the fall or spring of the study.
  Interventions: Workplace Wellness Program, Biometric Screening/HRA - No compensation, Wellness Activities - low compensation
  Interventions: Behavioral: Workplace Wellness Program; Behavioral: Biometric Screening/HRA - No Compensation; Behavioral: Wellness Activities - Low Compensation
- A75 (Experimental): Group A75 is offered no compensation for completing a biometric screening and HRA, and high compensation for each completed wellness course in the fall or spring of the study.
  Interventions: Workplace Wellness Program, Biometric Screening/HRA - No compensation, Wellness Activities - high compensation
  Interventions: Behavioral: Workplace Wellness Program; Behavioral: Biometric Screening/HRA - No Compensation; Behavioral: Wellness Activities - High Compensation
- B25 (Experimental): Group B25 is offered moderate compensation for completing a biometric screening and HRA, and low compensation for each completed wellness course in the fall or spring of the study.
  Interventions: Workplace Wellness Program, Biometric Screening/HRA - moderate compensation, Wellness Activities - high compensation
  Interventions: Behavioral: Workplace Wellness Program; Behavioral: Biometric Screening/HRA - Moderate Compensation; Behavioral: Wellness Activities - Low Compensation
- B75 (Experimental): Group B75 is offered moderate compensation for completing a biometric screening and HRA, and high compensation for each completed wellness course in the fall or spring of the study.
  Interventions: Workplace Wellness Program, Biometric Screening/HRA - moderate compensation, Wellness Activities - high compensation
  Interventions: Behavioral: Workplace Wellness Program; Behavioral: Biometric Screening/HRA - Moderate Compensation; Behavioral: Wellness Activities - High Compensation
- C25 (Experimental): Group C25 is offered high compensation for completing a biometric screening and HRA, and low compensation for each completed wellness course in the fall or spring of the study.
  Interventions: Workplace Wellness Program, Biometric Screening/HRA - high compensation, Wellness Activities - high compensation
  Interventions: Behavioral: Workplace Wellness Program; Behavioral: Biometric Screening/HRA - High Compensation; Behavioral: Wellness Activities - Low Compensation
- C75 (Experimental): Group C75 is offered high compensation for completing a biometric screening and HRA, and high compensation for each completed wellness course in the fall or spring of the study.
  Interventions: Workplace Wellness Program, Biometric Screening/HRA - high compensation Wellness Activities - high compensation
  Interventions: Behavioral: Workplace Wellness Program; Behavioral: Biometric Screening/HRA - High Compensation; Behavioral: Wellness Activities - High Compensation

INTERVENTIONS:
Behavioral: Workplace Wellness Program — Treatment group members will then be offered the opportunity to participate in a biometric screening and health risk assessment (biometric screening + HRA), and -- conditional on completing an biometric screening + HRA -- up to two, semester-long wellness programs. Treatment group members will be offered varying levels of cash reward for completing the biometric screening + HRA (none, moderate, high), and an additional cash reward for completing each wellness activity (low, high), for a total of 6 treatment cells. Follow-up surveys and biometric screenings will be administered one year later, among a subset of control and treatment group members.
  Other Names: Biometric Screening; Health Risk Assessment; Wellness Course
  Arms: A25; A75; B25; B75; C25; C75
Behavioral: Biometric Screening/HRA - No Compensation — The biometric test will measure: (1) anthropometrics such as height, weight, and waist circumference (to assess obesity and overweight status); (2) resting blood pressure (to assess hypertension); (3) blood glucose (to assess diabetes risk); and (4) total, LDL, and HDL cholesterol levels, total cholesterol ratio, and triglycerides (to assess risk of cardiovascular disease). The HRA is a survey designed to identify areas of health improvement, by asking a series of questions related to wellness, health status, nutrition, healthy activities, desire to improve health, preventative health measures. The HRA is also pre-populated with biometric information from the screening. Upon completion, participants are given customized feedback on areas of improvement. No compensation for completion.
  Arms: A25; A75
Behavioral: Biometric Screening/HRA - Moderate Compensation — The biometric test will measure: (1) anthropometrics such as height, weight, & waist circumference (to assess obesity and overweight status); (2) resting blood pressure (to assess hypertension); (3) blood glucose (to assess diabetes risk); & (4) total, LDL, and HDL cholesterol levels, total cholesterol ratio, and triglycerides (to assess risk of cardiovascular disease). The HRA is a survey designed to identify areas of health improvement, by asking a series of questions related to wellness, health status, nutrition, healthy activities, desire to improve health, preventative health measures. The HRA is also pre-populated with biometric information from the screening. Upon completion, participants are given customized feedback on areas of improvement. Moderate compensation for completion.
  Arms: B25; B75
Behavioral: Biometric Screening/HRA - High Compensation — The biometric test will measure: (1) anthropometrics such as height, weight, and waist circumference (to assess obesity and overweight status); (2) resting blood pressure (to assess hypertension); (3) blood glucose (to assess diabetes risk); and (4) total, LDL, and HDL cholesterol levels, total cholesterol ratio, and triglycerides (to assess risk of cardiovascular disease). The HRA is a survey designed to identify areas of health improvement, by asking a series of questions related to wellness, health status, nutrition, healthy activities, desire to improve health, preventative health measures. The HRA is also pre-populated with biometric information from the screening. Upon completion, participants are given customized feedback on areas of improvement. High compensation for completion.
  Arms: C25; C75
Behavioral: Wellness Activities - Low Compensation — Courses are designed by the UI Wellness Center and include an Active Living class; self-paced online health challenges in physical activity, weight management, and healthy eating; a weight management class; a tobacco cessation hotline; a stress management class; a Tai Chi class; and a chronic disease management class. Low compensation for each class.
  Arms: A25; B25; C25
Behavioral: Wellness Activities - High Compensation — Courses are designed by the UI Wellness Center and include an Active Living class; self-paced online health challenges in physical activity, weight management, and healthy eating; a weight management class; a tobacco cessation hotline; a stress management class; a Tai Chi class; and a chronic disease management class. High compensation for each class.
  Arms: A75; B75; C75

SUMMARY:
Workplace wellness programs have become a $6 billion industry and are widely touted as a way to improve employee well-being, reduce health care costs by promoting prevention, and increase workplace productivity. Yet, there is little rigorous evidence available to support these claims, partly because the voluntary nature of these programs means that participants may differ from nonparticipants for reasons unrelated to the causal effects of the wellness program. The investigators will implement a randomized control trial to identify the effects of incentives on wellness program participation, produce causal estimates of the effect of wellness programs on health outcomes, determine what kinds of employees benefit from wellness programs the most, and test for the presence of peer effects in wellness participation.

ELIGIBILITY:
Inclusion Criteria:

* Benefits eligible employees at UIUC. Physically located on UIUC campus, not terminated, eligible for benefits.

Exclusion Criteria:

* Members of the research team, employees directly involved with the approval or implementation of the study, family members of the research team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4834 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Wellness Program participation | First year of study
  Completion of biometric screening, HRA, wellness activities
Wellness Program participation | Second year of study
  Completion of biometric screening, HRA, wellness activities
Selection into treatment by baseline health spending | 13 months prior to study
  The investigators will compare the average observable characteristics of participants, relative to treatment non-participants. Average monthly spending prior to the intervention is measured via administrative health claims data.
Selection into treatment by self-reported health | Baseline measure
  The investigators will compare the average observable characteristics of participants, relative to treatment non-participants. Self-reported health is measured as excellent, good, average, or poor.
Selection into treatment by gender | Baseline measure
  The investigators will compare the average observable characteristics of participants, relative to treatment non-participants. Gender is measured in administrative HR records.
Selection into treatment by Age | Baseline measure
  The investigators will compare the average observable characteristics of participants, relative to treatment non-participants. Age is grouped into three categories: younger than 37, age 37 to 49, age 50 or higher.
Selection into treatment by race | Baseline measure
  The investigators will compare the average observable characteristics of participants, relative to treatment non-participants. Race is measure via administrative HR records, as white or nonwhite.
Selection into treatment by salary quartile | Baseline measure
  The investigators will compare the average observable characteristics of participants, relative to treatment non-participants. Salary, measured by administrative HR records, is coded into 1st, 2nd, 3rd, and 4th quartile.
Selection into treatment by self-reported health utilization | Baseline measure
  The investigators will compare the average observable characteristics of participants, relative to treatment non-participants. Health care utilization is measured by survey, with yes/no variable for: ever having been screened, prescription drug use, physician/ER visit in prior year, hospital visit in the past year.
Selection into treatment by smoking status | Baseline measure
  The investigators will compare the average observable characteristics of participants, relative to treatment non-participants. Smoking status is measured via survey, with yes/no variables for: current smoker of cigarettes, current smoker of other product, former smoker, never smoker.
Selection into treatment by chronic condition | Baseline measure
  The investigators will compare the average observable characteristics of participants, relative to treatment non-participants. Chronic condition is measured via baseline survey, and coded as a yes/no variable.
Health Insurance Spending | 12 months and 24-30 months following study
  Spending as measured in health insurance claims data
Employment and Productivity | 12 months and 24-30 months following study
  Promotion, job termination, sick leave, attitude toward management, index of these variables
Health Status and Behaviors | 12 months and 24-30 months following study
  Marathon participation, gym visits, health screening
Height | 1 year following study, 2 years following study
  Biometric health measures collected one year after study. Height is measured in feet and inches.
Weight | 1 year following study, 2 years following study
  Biometric health measures collected one year after study. Weight is measured in pounds and ounces.
Waist circumference | 1 year following study, 2 years following study
  Biometric health measures collected one year after study. Circumference is measured in inches.
Resting blood pressure | 1 year following study, 2 years following study
  Biometric health measures collected one year after study. Blood pressure is measured in mm Hg.
Blood glucose | 1 year following study, 2 years following study
  Biometric health measures collected one year after study. Blood glucose is measured in mg/dL.
Cholesterol levels | 1 year following study, 2 years following study
  Biometric health measures collected one year after study. Cholesterol is measured mg/dL. We measure lipids: LDL, HDL, and triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Jones, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Our study will collect detailed data on human subjects and perform several analyses using these data. These data will include self-reported survey data, biometric data, employer administrative data, and health care insurance claims data. Because our data are confidential and include protected health information, we can only share a de-identified version of the data. A statement is included on the study's informed consent form to secure participant's consent to make the de-identified data available to outside researchers. We will also provide replication code that will allow individuals to replicate all of our results. The public use version of our data and replication code for our analyses will be posted publicly on our study's website, which will be hosted at www.nber.org, as well as on the PI's websites.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available by July 2020, and will be available indefinitely.
Access Criteria: De-identified data, not linked across outcomes, will be available to download publicly. De-identified data, linked across outcomes, which is necessary for replication, will be available via a secure computer terminal at the National Bureau of Economic Research.
URL: http://www.nber.org/workplacewellness/downloads/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT03164330/Prot_SAP_000.pdf